CLINICAL TRIAL: NCT04092374
Title: Sternal Fracture Fixation by Locking Compression Plates (LCP) System
Brief Title: Assiut University Heart Hospital
Acronym: aun
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Ahmed Hosny, Resident Surgeon, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutUniv
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Sternal Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Case arm (Experimental)
  Interventions: Procedure: Locking compression plates

INTERVENTIONS:
Procedure: Locking compression plates — Fixation of sternal fracture using locking compression mechanism

SUMMARY:
It is interesting to examine this technique for sternal fracture fixation for more close-up assessment of post-operative pain using pain score, hospital stay and short-term complications. Investigators think that this approach will give the patient better post-operative results with less complications and excellent immediate relief with good quality of life, less post-operative pain and rapid return to normal life.

DETAILED DESCRIPTION:
Traumatic sternal fracture occurs due to direct anterior trauma to the chest or due to indirect trauma through flexion-compression of the spine. Trauma may lead to Type I manubri-sternal dislocation ( Corpi sterni displaced dorsally) or type II dislocation( corpi sterni is displaced ventrally) or it may lead to horizontal or longitudinal fractures.

Current management of such fractures includes conservative management as first line therapy. Correction Tape, plaster bandage, avoiding aggressive movement and analgesics are examples of conservative management. If the patient shows persistent pain, persistent displacement, instability, pressure over internal organs or vessels surgical reduction and fixation is indicated. However, there are no standard surgical approach for such fractures due to few numbers of studies and cases so it needs more investigations to establish evidence-based recommendations and standardization for these cases. Current surgical approaches include fixation using k-wires, cerclage wiring and more recently plates and screws.

Wiring fixation technique is the conventional technique used at our trauma centre. Investigators identified many complications from using wires as method of fixation. They include Sternal Wound Infection (SWI), sternal dehiscence, persistent pain and mal-alignment. They can be explained through the mechanism of fixation of plates. Loosening or tightening of wires twisting can lead to failure of function. In-complete burying of wires stump can lead to discomfort up-to painful sensation by the patient and may lead to sternal skin infection.

At contrast, Locking Compression Plates (LCP) system is a more recent technique used for sternal fractures fixation and is not thoroughly examined although it shows promising results at such cases. It does not depend on friction between bone and plates for fracture fixation which may fail at patients suffering from osteopenic bones or elder individuals. It depends on angle between screws and plates which is fixed showing long-term fixation over many years.

All of the previous made us interesting to examine this technique for sternal fracture fixation for more close-up assessment of post-operative pain using pain score, hospital stay and short-term complications. Investigators think that this approach will give the patient better post-operative results with less complications and excellent immediate relief with good quality of life, less post-operative pain and rapid return to normal life.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic sternal fractures
2. All patients of all ages and genders are included
3. All types of sternal fractures and manubri-sternal junction dislocation.

Exclusion Criteria:

1. All patient with Associated Injury Scale score of more than
2. Patients having their sternal fractures fixed using fixation approach other than LCP plates and screws.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Post operative pain: score | Early post operative period up to one week
  Pain score for post operative period in patients using locking compression plates.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university heart hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed K, Nady MA. Sternal reconstruction using locking compression plates (LCP): our experience in Egypt, a case series. J Cardiothorac Surg. 2020 Aug 21;15(1):224. doi: 10.1186/s13019-020-01266-0. PMID 32825827